CLINICAL TRIAL: NCT00397826
Title: Evaluation of the Effects of Simvastatin 40 Mg on Lipid Profiles and Specified Circulatory Parameters in Normotensive Hypercholesterolemia Patients(MK-0733-265)
Brief Title: Evaluation of the Effects of Simvastatin 40mg
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cardinal Tien Hospital (Other)
Responsible Party: Principal Investigator, Dong Feng Yeih, Attending Physician of Cardiology, Cardinal Tien Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0733-265
Record Dates: First submitted 2006-11-09; First posted 2006-11-10 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MK0733,simvastatin (Other): 20 patients with total cholesterol ≧ 240 mg/dL or LDL-C > 160 mg/dL for primary hypercholesterolemia; LDL-C ≧ 130 mg/dL for secondary hypercholesterolemia with identifiable risk factors will be enrolled into study to receive simvastatin 40 mg once daily for 12 weeks.
  Interventions: Drug: MK0733

INTERVENTIONS:
Drug: MK0733 — Duration of Treatment: 12 Weeks
  Other Names: simvastatin

SUMMARY:
To collect lipid-lowering response data with the use of simvastatin 40 mg tablet in patients with hypercholesterolemia.

DETAILED DESCRIPTION:
This is an open-label, prospective study to investigate lipid-lowering efficacy and sympathetic response of normotensive hypercholesterolemia patients after receiving simvastatin 40 mg once daily for 3 months.

The total duration of the study will be approximately 13 weeks, comprising of a 1-week (or 4 weeks?) screening period and a 12-week active treatment period. 20 hypercholesterolemia patients with normal blood pressure will be enrolled into treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient, >18 years of age
* Patients with hypercholesterolemia who meet the following lipid criteria:

  1. primary cholesterolemia: total cholesterol>=240 mg/dl or ldl-c >= 160 mg/dl
  2. secondary cholesterolemia (patients with cad, dm): ldl-c>=130 mg/dl
* The patient is willing to follow an NCEP therapeutic lifestyle changes (tlc) or similar cholesterol-lowering diet throughout the duration of the study

Exclusion Criteria:

* Congestive heart failure (NYHA class III or IV), uncontrolled cardiac arrhythmia, unstable angina
* Hypertension (based on the atp 3 guidelines)
* Taking potent lipid-lowering agents
* Unstable diabetes (hba1c >9%) or newly diagnosed (within 3 months), or a change in anti-diabetes medications within 3 months of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-01; Primary Completion 2006-01 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Total cholesterol, ldl-c, hdl-c, and triglycerides | after 12 weeks treatment

SECONDARY OUTCOMES:
Pulse wave velocity | after 12 weeks
Baroreflex sensitivity | after 12 weeks treatment
Serum nitrite, nitrate and urine c-gmp levels after 12 weeks treatment | after 12 weeks treatment

CONTACTS AND LOCATIONS:
Overall Officials: Dong Feng Yeih, MD,Phd, Principal Investigator — Cardinal Tiem Hospital

IPD SHARING:
Plan to Share IPD: No